CLINICAL TRIAL: NCT00701779
Title: Dutasteride (0.5mg) Once Daily for One Year and Tamsulosin (0.4mg) Once Daily for 3 Months, Followed by Counseling on Flex Dose Tamsulosin as Needed on Improvement of Symptoms and Outcome in Men With Moderate to Severe Symptomatic BPH
Brief Title: Dutasteride and Flex Dose of Tamsulosin on as Needed Basis, to Treat Benign Prostatic Hyperplasia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Siami, Paul F., M.D. (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Paul F. Siami, MD, Medical Director, Research Institute of Deaconess Clinic, Siami, Paul F., M.D.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Siami104907
Record Dates: First submitted 2008-06-17; First posted 2008-06-19 (Estimated); Results first posted 2015-01-01 (Estimated); Last update posted 2018-11-02 (Actual); Status verified 2018-11

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Benign Prostatic Hyperplasia; Dutasteride; Tamsulosin
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Tamsulosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dutasteride (Experimental): Dutasteride 0.5mg once daily for one year and tamsulosin 0.4mg administered once daily for 3 months, followed by counseling on flexible dosing of tamsulosin on an as needed basis.
  Subjects will self-administer the study medication once daily for up to 52 weeks (1 year). Subjects will return to the clinic at 13 week intervals during the treatment period. At each scheduled clinic visit (3, 6, and 9 months), the subjects will be counseled on withdrawal of Tamsulosin. The total study duration for each subject will be up to 52 weeks.
  Interventions: Drug: Tamsulosin

INTERVENTIONS:
Drug: Tamsulosin — Dutasteride 0.5mg once daily for one year and tamsulosin 0.4mg administered once daily for 3 months, followed by counseling on flexible dosing of tamsulosin on an as needed basis.
  Other Names: Flomax

SUMMARY:
This study will investigate the efficacy and safety of treatment with Dutasteride (0.5mg), administered once daily for one year in combination with Tamsulosin (0.4mg), administered once daily for 3 months, followed by counseling on flexible dosing of Tamsulosin on an as needed basis, on the improvement of symptoms and clinical outcome in men with moderate to severe symptomatic benign prostatic hyperplasia (BPH). At each scheduled visit (3, 6, and 9 months), the subject will be counseled on withdrawal of Tamsulosin. After randomization, study visits are every 13 weeks for up to 52 Weeks. (Including Screening, (up to 7 clinic visits)

DETAILED DESCRIPTION:
This study will investigate the efficacy and safety of treatment with Dutasteride (0.5mg), administered once daily for one year in combination with Tamsulosin (0.4mg), administered once daily for 3 months, followed by counseling on flexible dosing of Tamsulosin on an as needed basis, on the improvement of symptoms and clinical outcome in men with moderate to severe symptomatic benign prostatic hyperplasia (BPH). At each scheduled visit (3, 6, and 9 months), the subject will be counseled on withdrawal of Tamsulosin.

A recently published, landmark study (MTOPS - Medical Therapy of Prostatic Symptoms), co-sponsored by the National Institute of Health and the National Institute of Diabetes, Digestive and Kidney Diseases (NIH-NIDDK), demonstrated that, in selected patients, combination therapy with Doxazosin and Finasteride provided additive symptomatic improvements, reduced the risk of acute urinary retention (AUR) and surgical intervention, and was a more effective treatment for reduction in the overall risk of BPH clinical progression.

The aim of this proposed combination study, in a population of patients at high risk of BPH clinical progression, is to investigate whether combination therapy with Dutasteride and Tamsulosin with the subsequent withdrawal of Tamsulosin can maintain superior symptom improvement. At each scheduled visit (3, 6, and 9 months), the subject will be counseled on withdrawal of Tamsulosin. We hypothesize that patients may start with a combination of Dutasteride and Tamsulosin and eventually may be able to eliminate the use of Tamsulosin and maintain acceptable urinary symptoms on Dutasteride alone.

ELIGIBILITY:
Inclusion Criteria:

1. Male ≥50 yrs
2. Diagnosed BPH by medical history and physical examination, including a digital rectal examination
3. International Prostate Symptom Score ≥12 points at Screening
4. Prostate volume ≥30cc (by transrectal ultrasonography; TRUS)
5. Total serum Prostate Specific Antigen ≥1.5 ng/mL at Screening
6. Maximum flow rate ≥5 mL/sec and ≤15 mL/sec and minimum voided volume of ≥125 mL at Screening (based on two voids)
7. Able to give written informed consent and comply with study procedures
8. Literate in English language with the ability to read, comprehend, and record information on the IPSS, BII, and PPSM questionnaires
9. Able to swallow and retain oral medication
10. Able to participate for study duration

Exclusion Criteria:

1. Total serum PSA >10.0 ng/mL at Screening. Patients with total serum PSA >10.0 ng/mL may be acceptable for inclusion if the PSA elevation is thought to be due to BPH and not prostate cancer (by TRUS and biopsies showing no evidence of prostate cancer).
2. History or evidence of prostate cancer
3. Previous prostatic surgery or other invasive procedures to treat BPH
4. History of flexible/rigid cystoscopy or other instrumentation of the urethra within 7 days prior to Screening. Catheterization (<10F) is acceptable with no time restriction.
5. History of AUR within 3 months prior to Screening
6. Post-void residual volume >250mL (suprapubic ultrasound) at Screening
7. Any causes other than BPH, which may in the judgment of the investigator, result in urinary symptoms or changes in flow rate
8. History of breast cancer or clinical breast examination finding of unclear origin or suggestive of malignancy
9. Use of 5 alpha-reductase inhibitor, any drugs with antiandrogenic properties, or drugs noted for gynecomastia effects, within past 6 months and throughout the study. Previous use of AVODART within 12 months of the baseline or historical TRUS. Chronic use of Metronidazole is prohibited.
10. Concurrent use of anabolic steroids
11. Use of phytotherapy for BPH within 2 weeks of Screening
12. Use of any alpha-adrenoreceptor blockers within 2 weeks of Screening
13. Use of any alpha-adrenoreceptor agonists, anticholinergics or cholinergics within 48 hours prior to all uroflowmetry assessments.
14. Hypersensitivity to any alpha-/beta- adrenoreceptor blocker or 5-alpha-reductase inhibitor, or other chemically-related drugs.
15. Concurrent use of drugs known or thought to interaction with Tamsulosin.
16. History of hepatic impairment, abnormal liver function at Screening, History of renal insufficiency, serum creatinine >1.5 times the upper limit

18. history of malignancies other than basal cell carcinoma or squamous cell carcinoma of the skin within the past 2 years.

19. History of any illness the investigator might confound the results of the study or poses additional risk to the patient.

20. Any unstable, serious co-existing medical condition(s) 21. History of postural hypotension, dizziness, vertigo, or any other signs and symptoms of orthostasis.

22. History of 'first dose' hypotensive episode on initiation of alpha-l-adrenoreceptor antagonist therapy.

23. History of unsuccessful treatment with finasteride or Dutasteride 24. History or current drug or alcohol abuse within the previous 12 months. 25. Participation in any investigational or marketed drug trial within 30 days (or 5 half-lives whichever is the longer) preceding Screening and/or during the course of this study.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2005-09; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul F Siami, MD, Principal Investigator — Deaconess Clinic Research Institute
Locations (1):
- Research Institute of Deaconess Clinic, Evansville, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Medical Clinic
Pre-assignment Details: The population of subjects will be the 'Intent-toTreat' population.
Groups:
- Dutasteride: Dutasteride 0.5mg once daily for one year and tamsulosin 0.4mg administered once daily for 3 months, followed by counseling on flexible dosing of tamsulosin on an as needed basis.
  Subjects will self-administer the study medication once daily for up to 52 weeks (1 year). Subjects will return to the clinic at 13 week intervals during the treatment period. At each scheduled clinic visit (3, 6, and 9 months), the subjects will be counseled on withdrawal of Tamsulosin. The total study duration for each subject will be up to 52 weeks.
  Tamsulosin: Dutasteride 0.5mg once daily for one year and tamsulosin 0.4mg administered once daily for 3 months, followed by counseling on flexible dosing of tamsulosin on an as needed basis.
Period: Overall Study
Arm/Group | Dutasteride
Started | 63
3 Month | 60
6 Month | 58
9 Month | 56
12 Month | 54
Completed | 54
Not Completed | 9
Not completed — Adverse Event | 6
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: Enrollment of ~ 60 subjects will allow the proportion of subjects able to discontinue Tamsulosin, (assuming 50% able to discontinue), usage within 13% using a 95% confidence interval.
  Assuming 75% of the subjects are able to discontinue Tamsulosin, the proportion of subjects can be estimated to within 11% using a 95% confidence interval.
Arm/Group | Dutasteride
Number analyzed (Participants) | 54
Age, Customized [Mean (Standard Deviation); unit: years] | 66.63 (8.50)
Sex/Gender, Customized [Number; unit: participants]
  Male | 54
International Prostate Symptom Score (IPSS) [Mean (Standard Deviation); unit: units on a scale] — Questionnaire consisting of seven symptom scores: incomplete emptying, frequency, intermittency, urgency, weak stream, straining, and nocturia. Symptoms are scored on a 5 point scale with 0 representing absence of symptoms and 5 representing the most severe presentation of a symptom.
  Total range is from 0-35. The scores are evaluated as such:
  0-7: Mild 8-19: Moderate 20-35: Severe
  units on a scale | 19.80 (5.86)
Peak Flow Rate [Mean (Standard Deviation); unit: ml/sec] | 10.14 (2.64)
Prostate Specific Antigen [Mean (Standard Deviation); unit: ng/mL] | 4.70 (3.01)
Prostate Volume [Mean (Standard Deviation); unit: cc] | 57.61 (22.83)
Post-Void Residual Volume [Mean (Standard Deviation); unit: ml] | 82.33 (58.36)
Benign Prostatic Hyperplasia Impact Index (BII) [Mean (Standard Deviation); unit: units on a scale] — Benign Prostatic Hyperplasia Impact Index asked the following:
  1. Over the past month, how much physical discomfort did any urinary problems cause you? (0-3)
  2. Over the past month, how much did you worry about yoru health because of any urinary problems? (0-3)
  3. Overall, how bothersome has any trouble with urination been during the past month? (0-3)
  4. Over the past month, how much of the time has any urinary problem kept you from doing the kinds of things you usually do? (0-4) 0 indicates no symptoms, high values indicate high frequency of symptoms.
  Total symptom score range 0-13.
  units on a scale | 6.31 (3.11)

OUTCOME MEASURES:

1. Primary Outcome: International Prostate Symptom Score
Description: Reported mean total IPSS values from end of study (12 month visit) to assess efficacy of starting with combination treatment with Dutasteride for one year and Tamsulosin for 3 months with subsequent as needed use of Tamsulosin in providing superior symptomatic improvement to BPH patients.
  Questionnaire consisting of seven symptom scores: incomplete emptying, frequency, intermittency, urgency, weak stream, straining, and nocturia. Symptoms are scored on a 5 point scale with 0 representing absence of symptoms and 5 representing the most severe presentation of a symptom.
  Total range is from 0-35. The scores are evaluated as such:
  0-7: Mild 8-19: Moderate 20-35: Severe
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dutasteride
Number analyzed (Participants) | 54
units on a scale | 11.31 (6.48)

2. Primary Outcome: Peak Flow Rate (QMax)
Description: Peak flow rate recorded at final study visit (12 month) to assess efficacy of starting with combination treatment with Dutasteride for one year and Tamsulosin for 3 months with subsequent as needed use of Tamsulosin in providing superior symptomatic improvement to BPH patients.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: ml/sec
Arm/Group | Dutasteride
Number analyzed (Participants) | 54
ml/sec | 20.43 (38.68)

3. Primary Outcome: Benign Prostate Hyperplasia Impact Index
Description: Benign prostate hyperplasia Impact Index obtained at final study visit (12 month) to assess efficacy of starting with combination treatment with Dutasteride for one year and Tamsulosin for 3 months with subsequent as needed use of Tamsulosin in providing superior symptomatic improvement to BPH patients.
  Benign Prostatic Hyperplasia Impact Index asked the following:
  1. Over the past month, how much physical discomfort did any urinary problems cause you? (0-3)
  2. Over the past month, how much did you worry about yoru health because of any urinary problems? (0-3)
  3. Overall, how bothersome has any trouble with urination been during the past month? (0-3)
  4. Over the past month, how much of the time has any urinary problem kept you from doing the kinds of things you usually do? (0-4) 0 indicates no symptoms, high values indicate high frequency of symptoms. Total symptom score range 0-13.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dutasteride
Number analyzed (Participants) | 54
units on a scale | 3.28 (2.81)

4. Primary Outcome: Post-void Residual Volume
Description: Post-void residual volume taken at final study visit (12 month) to assess efficacy of starting with combination treatment with Dutasteride for one year and Tamsulosin for 3 months with subsequent as needed use of Tamsulosin in providing superior symptomatic improvement to BPH patients.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Dutasteride
Number analyzed (Participants) | 54
mL | 87.19 (83.47)

5. Primary Outcome: Prostate Specific Antigen
Description: Prostate Specific Antigen (PSA) taken at final study visit (12 month) to assess efficacy of starting with combination treatment with Dutasteride for one year and Tamsulosin for 3 months with subsequent as needed use of Tamsulosin in providing superior symptomatic improvement to BPH patients.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Dutasteride
Number analyzed (Participants) | 54
ng/mL | 1.91 (1.52)

6. Secondary Outcome: Health Outcome Measures
Description: Number of participants who are able to subsequently reduce or discontinue Tamsulosin usage after starting with combination therapy with Dutasteride and Tamsulosin while still maintaining the same degree of improvement in lower urinary tract symptoms
Time Frame: 13 months
Measure: Count of Participants; unit: Participants
Arm/Group | Dutasteride
Number analyzed (Participants) | 54
Participants | 31

7. Secondary Outcome: Safety and Tolerability
Description: To assess safety and tolerability of starting with combination therapy with Dutasteride and Tamsulosin and subsequent elimination of Tamsulosin. Evaluating number of reported adverse events designated as possibly or probably study-drug related.
Time Frame: 13 months
Measure: Number; unit: adverse events
Arm/Group | Dutasteride
Number analyzed (Participants) | 54
adverse events | 27

8. Secondary Outcome: Economic Impact
Description: Annual financial cost per participant starting with combination therapy with Dutasteride and Tamsulosin with subsequent withdrawal of Tamsulosin.
Time Frame: 13 months
Measure: Mean (Standard Deviation); unit: US dollars
Arm/Group | Dutasteride
Number analyzed (Participants) | 54
US dollars | 643.99 (306.91)

9. Secondary Outcome: Number of Participants With a Reduction of AUR and BPH-related Surgery
Description: To assess efficacy of starting with combination treatment with Dutasteride for one year and Tamsulosin for 3 months with subsequent as needed use of Tamsulosin in providing superior improvement in the clinical outcomes of AUR or BPH-related prostatic surgery to BPH patients.
Time Frame: 13 months
Measure: Count of Participants; unit: Participants
Arm/Group | Dutasteride
Number analyzed (Participants) | 54
Participants | 54

ADVERSE EVENTS:
Arm/Group | Dutasteride
Serious Adverse Events (participants affected / at risk) | 6/63
Other Adverse Events (participants affected / at risk) | 27/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dutasteride (N=63)
Chest Pain (Cardiac disorders) | 3 (3)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Cerebrovascular Accident (Vascular disorders) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 1 (1)
Peripheral Vascular Disease (Vascular disorders) | 1 (1)
Acute Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Right Lower Lobe
Osteoarthritis worsening (Musculoskeletal and connective tissue disorders) | 1 (1) — Left knee
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dutasteride (N=63)
Fatigue (General disorders) | 3 (3)
Lower Abdominal Pain (Gastrointestinal disorders) | 4 (4)
Back Pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Sinus Infection (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Laceration (Injury, poisoning and procedural complications) | 3 (3) — Hand, arm, finger
Rash (Skin and subcutaneous tissue disorders) | 4 (4) — calf(s), groin, arm(s), abdomen, neck
Retrograde Ejaculation (Reproductive system and breast disorders) | 8 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No